CLINICAL TRIAL: NCT07092891
Title: Early Detection of Supraclavicular Brachial Plexus Block Failure Using Infrared Thermography and Perfusion Index: Randomized Double-Blind Controlled Study
Brief Title: Early Detection of Supraclavicular Brachial Plexus Block Failure Using Infrared Thermography and Perfusion Index
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Tarek Ashraf Ibrahim Abd Al-Hafiz, resident doctor at Assiut University hospital, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Brachial Plexus Block Failure
Record Dates: First submitted 2025-07-15; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Regional Anaesthsia; Brachial Plexus Blocks
Keywords: Brachial Plexus Blocks; Regional Anaesthesia
MeSH Terms: interventions — Bupivacaine; Ultrasonography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supraclavicular Brachial Plexus Block with Thermographic and Perfusion Monitoring (Experimental): Participants will receive an ultrasound-guided supraclavicular brachial plexus block using 30 mL of 0.5% bupivacaine for upper limb surgery. Infrared thermography and perfusion index measurements will be recorded at baseline, and at 5, 10, and 15 minutes post-block to detect early physiological changes. Clinical assessment of sensory and motor block will be performed at 20 minutes post-injection using standardized testing. The goal is to evaluate the predictive accuracy of these non-invasive measures in detecting block success or failure.
  Interventions: Procedure: Ultrasound-Guided Supraclavicular Block; Drug: Bupivacaine Hydrochloride 0.5 % Injectable Solution; Device: Ultrasound; Device: Infrared Thermography Camera; Device: Pulse Oximeter

INTERVENTIONS:
Procedure: Ultrasound-Guided Supraclavicular Block — Ultrasound-guided supraclavicular brachial plexus block using a high-frequency linear ultrasound probe-real-time visualization of the brachial plexus for precise anesthetic delivery.
Drug: Bupivacaine Hydrochloride 0.5 % Injectable Solution — 30 mL used for supraclavicular brachial plexus block
Device: Ultrasound — Imaging for block placement
Device: Infrared Thermography Camera — Skin temperature monitoring
Device: Pulse Oximeter — Perfusion Index monitoring

SUMMARY:
Successful peripheral nerve blockade is fundamental to modern regional anesthesia, particularly for upper limb surgeries. Ensuring the efficacy of a nerve block early in the perioperative period is critical, as delayed recognition of block failure may lead to intraoperative pain, the need for additional sedation or general anesthesia, and overall poorer patient outcomes. Conventional methods for assessing block success, such as sensory testing with pinprick or cold stimuli and motor assessment using strength scales, require patient cooperation and often take 15-30 minutes to yield definitive results. These delays are especially limiting in fast-paced surgical environments or when early decisions regarding anesthesia management are necessary.

Emerging non-invasive monitoring technologies offer promising alternatives for the early, objective assessment of block efficacy. Infrared Thermography (IRT) measures skin surface temperature, which increases due to sympathetic nerve blockade-induced vasodilation.

DETAILED DESCRIPTION:
Successful peripheral nerve blockade is fundamental to modern regional anesthesia, particularly for upper limb surgeries. Ensuring the efficacy of a nerve block early in the perioperative period is critical, as delayed recognition of block failure may lead to intraoperative pain, the need for additional sedation or general anesthesia, and overall poorer patient outcomes. Conventional methods for assessing block success, such as sensory testing with pinprick or cold stimuli and motor assessment using strength scales, require patient cooperation and often take 15-30 minutes to yield definitive results. These delays are especially limiting in fast-paced surgical environments or when early decisions regarding anesthesia management are necessary.

Emerging non-invasive monitoring technologies offer promising alternatives for early, objective assessment of block efficacy. Infrared Thermography (IRT) measures skin surface temperature, which increases with sympathetic nerve blockade-induced vasodilation. Perfusion Index (PI), derived from pulse oximetry, reflects peripheral perfusion and also rises as vascular tone decreases following a successful nerve block. Both IRT and PI provide quantifiable, real-time physiological markers of sympathetic and circulatory changes that precede full sensory or motor blockade. Although several studies support their individual utility, there is limited evidence on their combined predictive value or their integration into routine clinical practice. Further investigation is needed to validate their role in enhancing the accuracy and timeliness of block assessment.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-70 years
* ASA Physical Status I-III

Exclusion Criteria:

* General

  * Coagulopathy
  * Allergy to local anesthetics
* Special

  * Neurological deficits in the affected limb
  * Peripheral vascular disease or Raynaud's phenomenon
  * Infections or skin lesions at the site of injection
  * Use of a tourniquet

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Skin Temperature (°C) Measured by Infrared Thermography From Baseline to 10 Minutes Post-block. | Baseline, 5, and 10 minutes post-injection
  Mean change in skin temperature on the operative limb captured using infrared thermography at defined time points.
Change in Perfusion Index From Baseline to 10 Minutes Post-block | Baseline, 5, and 10 minutes post-injection
  PI measured via pulse oximeter; change calculated as ratio to baseline values.

SECONDARY OUTCOMES:
Correlation Between Changes in Skin Temperature and Perfusion Index With Sensory and Motor Block Scores at 20 Minutes | 20 minutes post-injection
  Correlation between physiologic changes and clinical assessments of sensory and motor block success using pinprick/cold test and Modified Bromage Scale.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gamal M, Hasanin A, Adly N, Mostafa M, Yonis AM, Rady A, Abdallah NM, Ibrahim M, Elsayad M. Thermal Imaging to Predict Failed Supraclavicular Brachial Plexus Block: A Prospective Observational Study. Local Reg Anesth. 2023 Jun 9;16:71-80. doi: 10.2147/LRA.S406057. eCollection 2023. PMID 37323293
- [Background] Abdelnasser A, Abdelhamid B, Elsonbaty A, Hasanin A, Rady A. Predicting successful supraclavicular brachial plexus block using pulse oximeter perfusion index. Br J Anaesth. 2017 Aug 1;119(2):276-280. doi: 10.1093/bja/aex166. PMID 28854539